CLINICAL TRIAL: NCT06462144
Title: An Exploartory Trial of IMPT-514, An Autologous Anti-CD19/20 CAR T Therapy in Participants With Active, Refractory Systemic Lupus Erythematosus, Anca-associated Vasculitis, and Idiopathic Inflammatory Myopathy
Brief Title: IMPT-514 in Systemic Lupus Erythematosus, Anca-associated Vasculitis, and Idiopathic Inflammatory Myopathy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The collaborating party has adjusted its R&D strategy and terminated the study.
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Lingyun Sun, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD17-01
Record Dates: First submitted 2024-06-04; First posted 2024-06-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE); ANCA Associated Vasculitis (AAV); Idiopathic Inflammatory Myopathy (IIM)
Keywords: CD19/CD20 CART
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): IMPT-514
  Interventions: Drug: IMPT-514 CART Cell Injection

INTERVENTIONS:
Drug: IMPT-514 CART Cell Injection — CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide.

SUMMARY:
This is an exploratory trial to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of a single dose of IMPT-514, an autologous, anti-CD19/CD20 CAR T therapy, administered as an intravenous (IV) infusion, in participants with B cell driven autoimmune diseases, including active, refractory Systemic Lupus Erythematosus (SLE), ANCA Associated Vasculitis (AAV), and Idiopathic Inflammatory Myopathy (IIM).

DETAILED DESCRIPTION:
This study will explore the safety of IMPT-514 and will include up to two dose levels, with up to 12 total expected dosed participants for each disease group of SLE, AAV, and IIM.

IMPT-514 treatment consists of a single infusion of CAR-transduced autologous T cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide. Individual participants will remain in the active post-treatment period for approximately 2 year from IMPT-415 administration.

ELIGIBILITY:
General Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Age 18 years of age or older and ≤75 years.
3. Weight > 35 kg at enrollment.
4. On stable background therapy (such as mycophenolate, cyclophosphamide, etc.) for autoimmune disease (SLE, AAV, IIM) with stable dose of immunosuppressants for at least 4 weeks prior to screening.

For SLE participants:

1. Diagnosis of SLE according to the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria or 2012 Systemic Lupus Collaborating Clinics (SLICC) criteria, including positive ANA >1:80 or positive anti-dsDNA.

For AAV participants:

1. Meets the diagnostic criteria for ANCA vasculitis in 2022 ACR/EULAR, including microscopic polyangiitis (MPA), granulomatous polyangiitis (GPA), and eosinophilic granulomatous polyangiitis (EGPA).

For IIM (Dermatomyositis, Anti-Synthetase Syndrome, and Immune-Mediated Necrotizing Myopathy) participants:

1. Diagnosis of probable or definite IIM with subgroup classification of dermatomyositis, or immune-mediated necrotizing myopathy (IMNM) subgroup of polymyositis.

Exclusion Criteria:

1. Any clinically significant underlying illness, other than systemic autoimmune disease (SLE, AAV, IIM), which would pose a safety risk or concern, as determined by the Investigator.
2. Rapidly progressive glomerulonephritis.
3. For SLE participants: Active central nervous system (CNS) lupus.
4. History of, or current significant neurologic disease.
5. History of allogeneic bone marrow or stem cell transplantation or solid organ transplantation (such as kidney, lung, heart transplant) or plans for such transplantation in future.
6. History of prior CAR T treatment, autologous or allogeneic.
7. Drug induced SLE, drug induced vasculitis or drug induced myopathy or myositis.
8. Any primary immunodeficiency.
9. History of, or current significant cardiovascular dysfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs), serious adverse events (SAE) and treatment-emergent adverse events (TEAEs). | 28 days from cell infusion

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The Affiliated Hospital Of Xuzhou Medical University, Xuzhou, Jiangsu
  - Zhongshan Hospital Fudan University., Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No